CLINICAL TRIAL: NCT03163979
Title: Individualized Precise Radiotherapy With the Guidance of Radiosensitivity: A Study on the Clinical Management Model of Locally Advanced Cervical Cancer
Brief Title: Individualized Precise Radiotherapy With the Guidance of Radiosensitivity of Locally Advanced Cervical Cancer
Acronym: PROGRAMMA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ke Gu, associate professor, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE2015645
Record Dates: First submitted 2017-04-17; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Cervical Cancer
Keywords: locally advanced cervical cancer; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PET/CT and Comet assay guided IMRT (Active Comparator): 18F-FDG PET/CT and Comet assay guide IMRT Based on FDG-PET/CT and comet analysis, higher doses of irradiation can be delivered to low sensitivity tumor region, so as to achieve individualized treatment.
  Interventions: Biological: 18F-FDG PET/CT and Comet assay guide IMRT
- PET/CT and Comet assay guided RapidArc (Active Comparator): 18F-FDG PET/CT and Comet assay guide RapidArc:
  1.A Rapid-Arc plan for cancer of the cervix uteri improved the sparing of organs at risk (OARs) with uncompromised target coverage. 2.Based on FDG-PET/CT and comet analysis, higher doses of irradiation can be delivered to low sensitivity tumor region, so as to achieve individualized treatment.
  Interventions: Biological: 18F-FDG PET/CT and Comet assay guide RapidArc
- RapidArc (Active Comparator): RapidArc:
  A maximum DR of 600 MU/min was set for comparing the 7f-IMRT treatment time. Two 360° coplanar arcs (one clockwise arc rotated from 181° to 179° and the other counter-clockwise arc rotated from 179° to 181°) sharing the same isocentre were used.
  Interventions: Biological: RapidArc
- 7f-IMRT (Sham Comparator): seventy-five patients received IMRT. The 7f-IMRT gantry angles were 0°, 51°, 102°, 153°, 204°, 255° and 306°, with 20 intensity levels and a dose rate of 400 monitor units (MU)/min. Doses were delivered using the step-and-shoot method.Conventional fractionation was used in all patients for a total dose 45-50.4 Gy with 6 MV high-energy photons.
  Interventions: Biological: 7f-IMRT

INTERVENTIONS:
Biological: 18F-FDG PET/CT and Comet assay guide RapidArc — 1.A Rapid-Arc plan for cancer of the cervix uteri improved the sparing of organs at risk (OARs) with uncompromised target coverage. 2.Based on FDG-PET/CT and comet analysis, higher doses of irradiation can be delivered to low sensitivity tumor region, so as to achieve individualized treatment.
  Arms: PET/CT and Comet assay guided RapidArc
Biological: 18F-FDG PET/CT and Comet assay guide IMRT — Based on FDG-PET/CT and comet analysis, higher doses of irradiation can be delivered to low sensitivity tumor region, so as to achieve individualized treatment.
  Arms: PET/CT and Comet assay guided IMRT
Biological: RapidArc — RapidArc:
  A maximum DR of 600 MU/min was set for comparing the 7f-IMRT treatment time. Two 360° coplanar arcs (one clockwise arc rotated from 181° to 179° and the other counter-clockwise arc rotated from 179° to 181°) sharing the same isocentre were used.
  Arms: RapidArc
Biological: 7f-IMRT — seventy-five patients received IMRT. The 7f-IMRT gantry angles were 0°, 51°, 102°, 153°, 204°, 255° and 306°, with 20 intensity levels and a dose rate of 400 monitor units (MU)/min. Doses were delivered using the step-and-shoot method.Conventional fractionation was used in all patients for a total dose 45-50.4 Gy with 6 MV high-energy photons.
  Arms: 7f-IMRT

SUMMARY:
Cisplatin-based chemoradiation (CCRT) has been considered as the standard care for patients with locally advanced cervical cancer (LACC). Nevertheless, increasingly more radio-resistant tumors still recur. IMRT including Rapid-Arc have obvious advantage in the dose distribution and organ protection, and positron emission tomography (PET) with F-18 fluorodeoxyglucose (FDG) and Comet analysis have good sensitivity for detecting sites and radiosensitivity of disease. These may be helpful to individualized CCRT of LACC.

Three hundred LACC patients are enrolled in the study, who were with FIGO stages IB2-IVA and had no para-aortic lymphadenopathy (>10 mm) assessed by PET-CT or MRI. All the patients received definitive radiotherapy consisting of external beam whole pelvic RT and HDR-ICBT. The cumulative linear quadratic equivalent dose (EQD2) was 70-75Gy prescribed at point A. Cisplatin 30 mg/m2 weekly was administered concurrently for 5 courses. 2-4 cycles TP (Taxol 135 mg/m2, D1 and DDP 25 mg/m2, D1-3) regimen sequential chemotherapy were performed if complete response (CR) not achieved according to magnetic resonance imaging (MRI) or PET-CT after CCRT. Hypothesis of the study is that CCRT and sequential chemotherapy is safe. Based on FDG-PET/CT and Comet assay, higher doses can be safely delivered individually to accurate tumor volume, while the doses to bladder and rectum are relative low. Comet and FDG-PET/CT-guided IMRT including RapidArc may improve survival in terms of time to progression (TTP), progression-free survival (PFS) and overall survival (OS) and less treatment-related toxicity. The data will be observed and analyzed.

DETAILED DESCRIPTION:
Cisplatin-based chemoradiation (CCRT) has been considered as the standard care for patients with locally advanced cervical cancer (LACC). Nevertheless, increasingly more radio-resistant tumors still recur. IMRT including Rapid-Arc have obvious advantage in the dose distribution and organ protection, and positron emission tomography (PET) with F-18 fluorodeoxyglucose (FDG) and Comet analysis have good sensitivity for detecting sites and radiosensitivity of disease. These may be helpful to individualized CCRT of LACC. IMRT including RapidArc could be considered as a treatment selection for LACC patients, and it aims to improve the degree of target coverage, to protect organ at risk (OARs) and healthy tissue sparing compared to other RT solutions and to reduce significantly the treatment time as to RapidArc. Several studies have indicated that FDG-PET/CT increases the accordance between biopsies and delineated tumor volume and has the potential to positively impact the course of treatment. The Comet assay is attractive as a potential clinical test of tumour radiosensitivity. During radiotherapy, accurately defining disease areas is critical to avoid unnecessary irradiation of normal tissue. Based on FDG-PET/CT and Comet assay, higher doses can be safely delivered individually to accurate tumor volume, while the doses to bladder and rectum are relative low.

Three hundred LACC patients are enrolled in the study, who were with FIGO stages IB2-IVA and had no para-aortic lymphadenopathy (>10 mm) assessed by PET-CT or MRI. All the patients received definitive radiotherapy consisting of external beam whole pelvic RT and HDR-ICBT. The cumulative linear quadratic equivalent dose (EQD2) was 70-75Gy prescribed at point A. Cisplatin 30 mg/m2 weekly was administered concurrently for 5 courses. 2-4 cycles TP (Taxol 135 mg/m2, D1 and DDP 25 mg/m2, D1-3) regimen sequential chemotherapy were performed if complete response (CR) not achieved according to magnetic resonance imaging (MRI) or PET-CT after CCRT. Hypothesis of the study is that CCRT and sequential chemotherapy is safe. Comet and FDG-PET/CT-guided IMRT including RapidArc may improve survival in terms of time to progression (TTP), progression-free survival (PFS) and overall survival (OS) and less treatment-related toxicity. The data will be observed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 18-70 years old;
2. Histology or cytology confirmed cervical squamous cell carcinomas;
3. 2009 FIGO stage includesⅠB2, ⅡA2, ⅡB-ⅣA;
4. Performance status(PS): 0-1;
5. Peripheral blood meet the following conditions: neutrophil count > 2.0 * 109/L, white blood cell count > 4.0 * 109/L, the platelet count > 100.0 * 109/L;
6. Liver and kidney function meet the following conditions: bilirubin < 1.5 mg/dl, AST and ALT < 2 times the upper limit of normal serum creatinine < 1.5 mg/dl, creatinine clearance > 50 ml/min;
7. Signed informed consent before treatment.

Exclusion Criteria:

1. There is no definite pathological diagnosis;
2. Clinical or imaging examination revealed distant metastases;
3. Pelvic had received radiotherapy;
4. Patients can't attend the study because of the associated with other diseases;
5. Patients can't sign the informed consent because of mental disorders, mental disorders;
6. Uncontrolled active infection;
7. No follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression-Free-Survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall survival
TTP | 3years
  Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-liang Ding, Study Chair — Health and Family Planning Commission of Jiangsu Province, China
Locations (1):
- Nanjing Medical University Affiliated Suzhou Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji S, Hu Q, Zhu J, Chen J, Chen Q, Liu Z, Shen C, Yang R, Sun H, Wu J, Gu K. Combined pretreatment with 18F-FDG PET/CT and Comet assay guides the concurrent chemoradiotherapy of locally advanced cervical cancer: study protocol for a randomized controlled trial. Trials. 2018 Aug 3;19(1):416. doi: 10.1186/s13063-018-2800-7. PMID 30075736